CLINICAL TRIAL: NCT00261638
Title: A Study of the Effect of Mental Health Promotion on Mental Health Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701123
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2005-12-05 (Estimated); Status verified 2005-10

CONDITIONS: Healthy
Keywords: Mental Health Promotion; Mental Health Index; Taiwan Mental Health Index scale; psychophysical health; education years over 9 years; normal people, especially joining Mental Health Foundation Promotions

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
"Health" includes physical and mental aspects. The evaluation of "Mental Health" contains four domains: psychophysical health, perceived security of the living world, meaning and worth of life, satisfaction of family-social interaction.

We have established a Taiwan Mental Health Index scale based on literature review and experts' opinions in 2002. The reliability and validity were assessed to be satisfactory. This TMHI scale has been applied in nation-wide mental health surveys of 2002, 2003, and 2004.

In order to evaluate the effect of mental health promotion activities, this research project will adopt this TMHI scale as the assessment tool. 300 people will be recruited for study after signing the informed consent. The general population sample of 1076 subjects recruited in 2004, will be as the comparison sample. The difference in 4 dimensions of MHI will be analyzed between these two study groups. The 300 study subjects will be subcategorized into two groups of low and high attendance groups. The difference in MHI between groups will also be statistically examined using independent t-test. The statistical signification is set at α=0.05.

This study result will be as the reference for setting up effective mental health promotion program for general public.

ELIGIBILITY:
Inclusion Criteria:

* Normal people
* education years over 9 years
* with reading ability

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-10; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University
Locations (1):
- Mental Health Foundation/ Wonderful Brain, Taipei, Taipei, Taiwan